CLINICAL TRIAL: NCT04123912
Title: Effect of Kinesio Taping and Functional Movement Power Training on Neuromuscular Performance, Motor Proficiency and Functional Independence in Children With Developmental Coordination Disorder: A Randomised Controlled Trial
Brief Title: Kinesio Taping and Physiotherapeutic Exercises for Children With DCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shirley S.M. Fong, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Developmental Coordination Disorder
MeSH Terms: conditions — Motor Skills Disorders | interventions — Jogging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT-FMPT group (Experimental)
  Interventions: Behavioral: Kinesio Taping - Functional Movement Power Training
- Control group (Placebo Comparator)
  Interventions: Behavioral: Jogging with placebo taping

INTERVENTIONS:
Behavioral: Kinesio Taping - Functional Movement Power Training — Subjects assigned to the Kinesio Taping - Functional Movement Power Training (KT-FMPT) group will receive FMPT concurrent with KT. The FMPT protocol was developed by the research team with reference to common physiotherapeutic exercises for children with motor disabilities.9 It comprises 5 functional movement exercises and 6 lower-limb power/resistance training exercises using weights or resistance bands.
  Arms: KT-FMPT group
Behavioral: Jogging with placebo taping — Subjects assigned to the control group will receive no FMPT or KT, but participate in a jogging intervention with placebo tape applied on their calf muscles and removed after the intervention.
  Arms: Control group

SUMMARY:
Aim: To investigate the effectiveness of a novel elastic taping-augmented functional movement power training (KT-FMPT) program in improving leg muscular performance, body balance, motor proficiency and functional independence in children with developmental coordination disorder (DCD).

Methodology: In this clinical trial, twenty children with DCD (aged 6-12) will be randomly assigned to either a KT-FMPT group or a placebo control group. Children in the KT-FMPT and control groups will receive elastic taping-augmented FMPT and general jogging exercise with non-elastic taping, respectively, for 12 weeks (2 hours/week). Major outcome measures: body balance and leg muscle activity will be measured via muscle sensors along with a force platform. Secondary outcome measures: leg muscle strength, motor proficiency and functional independence will be assessed by a digital dynamometer, the Movement Assessment Battery for Children-2 and Pediatric Evaluation of Disability Inventory, respectively (before- and after-intervention measurements).

Significance: The KT-FMPT group is predicted to display much better muscular and motor performances than the control group. This novel training program can be readily adopted in clinical, school, or home settings to improve functional independence in children with DCD, an outcome with positive socioeconomic implications. Moreover, study findings will inspire future research work in children with other childhood-onset disabilities.

ELIGIBILITY:
Inclusion Criteria:

* 6- to 12-years-old
* classified as DCD according to the Diagnostic and Statistical Manual of Mental Disorders V
* score < 5th percentile on the Movement Assessment Battery for Children, 2nd edition (MABC-2)
* total score < 46 on the DCD questionnaire (2007)
* attending a mainstream primary school with intelligence level within the normal range
* no KT or FMPT experience

Exclusion Criteria:

* any known congenital, cognitive, psychiatric, neurological, sensorimotor, musculoskeletal or cardiopulmonary disorder that may affect test performance
* receiving active rehabilitation treatment
* demonstrating excessive disruptive behaviour
* unable to follow instructions

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in leg muscle electromyographic activation onset latency time (in ms) | 0 and 3 months
  Electromyographic activation onset of leg muscles
Change in centre of pressure movement pathway in standing (in mm/cm) | 0 and 3 months
  Centre of pressure movement pathway in standing

SECONDARY OUTCOMES:
Change in lower-extremity maximum isometric muscle strength (in kg/N) | 0 and 3 months
  Maximum isometric leg muscle strength
Change in Movement Assessment Battery for Children-2 percentile score | 0 and 3 months
  Movement Assessment Battery for Children-2 percentile (motor proficiency)
Change in Pediatric Evaluation of Disability Inventory score | 0 and 3 months
  Pediatric Evaluation of Disability Inventory score (functional independence)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided